CLINICAL TRIAL: NCT00411086
Title: Single-Arm, Open-Label, Phase II Trial of Rituximab Plus Sargramostim for the Treatment of Newly Diagnosed Follicular B-Cell Lymphoma in Adults
Brief Title: Rituximab and GM-CSF in Treating Patients With Newly Diagnosed Follicular B-Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDA-2006-0260; P30CA016672 (NIH); MDA-2006-0260 (Other: UT MD Anderson Cancer Center); CDR0000521620 (Registry Identifier: NCI PDQ); NCI-2009-00187 (Registry Identifier: NCI CTRP); NCT00409474 (obsolete NCT alias)
Record Dates: First submitted 2006-12-11; First posted 2006-12-13 (Estimated); Results first posted 2017-12-05 (Actual); Last update posted 2017-12-05 (Actual); Status verified 2017-11

CONDITIONS: Lymphoma
Keywords: contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; stage I grade 1 follicular lymphoma; stage I grade 2 follicular lymphoma; stage I grade 3 follicular lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; Granulocyte-Macrophage Colony Stimulating Factor; GM-CSF; Rituximab; Rituxan
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular | interventions — Rituximab; sargramostim; Granulocyte-Macrophage Colony-Stimulating Factor; Colony-Stimulating Factors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Rituximab + GM-CSF (Experimental): Rituximab 375 mg/m^2 By Vein Weekly on Days 1, 8, 15, and 22. Sargramostim (GM-CSF) 250 mcg subcutaneously three times weekly for 8 weeks, starting at least 1 hour before first dose of rituximab.
  Interventions: Biological: Rituximab; Biological: Sargramostim (GM-CSF)

INTERVENTIONS:
Biological: Rituximab — 375 mg/m^2 By Vein Weekly on Days 1, 8, 15, and 22.
  Other Names: Rituxan
Biological: Sargramostim (GM-CSF) — 250 mcg subcutaneously three times weekly for 8 weeks, starting at least 1 hour before first dose of rituximab.
  Other Names: Granulyte; Leukene; Granulocyte-Macrophage Colony Stimulating Factor

SUMMARY:
RATIONALE: Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Colony-stimulating factors, such as GM-CSF, may increase the number of immune cells found in bone marrow or peripheral blood. Giving rituximab together with GM-CSF may be an effective treatment for follicular B-cell lymphoma.

PURPOSE: This phase II trial is studying the side effects and how well giving rituximab together with GM-CSF works in treating patients with newly diagnosed follicular B-cell lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety and efficacy of rituximab and sargramostim (GM-CSF), in terms of complete response at 12 weeks, in patients with newly diagnosed follicular B-cell lymphoma.

Secondary

* Determine the overall response rate in patients treated with this regimen.
* Determine the progression-free survival at 3 years in patients treated with this regimen.
* Determine the adverse event profile of this regimen in these patients.
* Determine the survival of patients treated with this regimen.
* Determine the effect of Fc gamma receptor polymorphism on response rate and time to progression in patients treated with this regimen.

OUTLINE: This is an open-label, multicenter study.

Patients receive rituximab IV on days 1, 8, 15, and 22 and sargramostim (GM-CSF) subcutaneously on days 1, 3, and 5. Treatment with GM-CSF repeats weekly for up to 8 weeks in the absence of disease progression or unacceptable toxicity.

Patients undergo blood collection at baseline for correlative laboratory studies of Fc-gamma receptor RIIIa 158 polymorphism.

After completion of study treatment, patients are followed every 3 months for 2 years and then every 6 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically confirmed newly diagnosed follicular B-cell lymphoma.
2. Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >/= 20 mm with conventional techniques or as >/= 10 mm with spiral CT scan.
3. Patients should not have received prior therapy of any kind for follicular B-cell lymphoma.
4. Age >/= 18 years. Because no dosing or adverse event data are currently available for the use of rituximab in combination with sargramostim in patients (males or females) <18 years of age, children are excluded from this study.
5. Eastern Cooperative Oncology (ECOG) performance status </= 2 (Karnofsky >/= 60%).
6. Patients must have normal organ and marrow function as defined below: - leukocytes >/= 3,000/microL; - absolute neutrophil count >/= 1,500/microL; - platelets >/= 100,000/microL; -total bilirubin within normal institutional limits; - AST(SGOT)/ALT(SGPT) </= 2.5 X institutional upper limit of normal; - creatinine within normal institutional limits OR - creatinine clearance >/= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
7. Hemoglobin >/= 8.0 gm/dL
8. The effects of rituximab and sargramostim on the developing human fetus at the recommended therapeutic doses are unknown. For this reason women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
9. Ability to understand and the willingness to sign an informed consent document.

Exclusion Criteria:

1. Prior therapy of any kind for follicular B-cell lymphoma.
2. Patients may not be receiving any other investigational agents.
3. Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
4. History of allergic reactions attributed to compounds of similar chemical or biologic composition to rituximab or other agents used in the study.
5. Rituximab is contraindicated in patients with known anaphylaxis or IgE-mediated hypersensitivity to murine proteins. Sargramostim is contraindicated in patients with excessive leukemic myeloid blasts, with known hypersensitivity to GM-CSF or yeast-derived components of the recombinant, and for concomitant (or within 24 hours ± of) uses with chemotherapy or radiotherapy.
6. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
7. Pregnant women are excluded from this study.
8. Patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy. Therefore, HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions.
9. Patients with evidence of active or prior infection of Hepatitis B are excluded. (Note: Persons vaccinated for Hepatitis B who have positive antibodies are not excluded).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-11; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Fowler, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Official Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: December 2006 and May 2009. All recruitment was done in medical clinics in participating Community Clinical Oncology Program sites.
Period: Overall Study
Arm/Group | Rituximab + GM-CSF
Started | 52
Completed | 52
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Rituximab + GM-CSF
Number analyzed (Participants) | 52
Age, Continuous [Median (Full Range); unit: years] | 57 [31 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 51
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 49
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 52

OUTCOME MEASURES:

1. Primary Outcome: Complete Response Rate
Description: Complete disappearance of all detectable clinical and radiographic evidence of disease and disappearance of all disease-related symptoms if present before therapy, and normalization of those biochemical abnormalities [e.g., lactate dehydrogenase (LDH)] definitely assignable to NHL.
  Response and progression evaluated using the International Criteria proposed in the Report of an International Workshop to Standardize Response Criteria for Non-Hodgkin's Lymphomas.
Time Frame: 12 weeks (3 months)
Population: Response includes unconfirmed CRs.
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab + GM-CSF
Number analyzed (Participants) | 52
percentage of participants | 23

2. Secondary Outcome: Median Progression-Free Survival (PFS)
Description: PFS is defined as the duration of time from start of treatment to time of progression; and, for PFS time calculated from chemo start date to progression date or death date, whichever happened first. Patients were censored at the last follow-up date if neither progression nor death occurred. Response and progression evaluated using the International Criteria proposed in the Report of an International Workshop to Standardize Response Criteria for Non-Hodgkin's Lymphomas. The Kaplan-Meier method was used for time-to-event analysis including PFS.
Time Frame: 3 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Rituximab + GM-CSF
Number analyzed (Participants) | 52
Months | 25 [15.3 to 59.9]

3. Secondary Outcome: Overall Response (OR) Rate
Description: OS defined as percentage of participants alive at a certain period following start of chemotherapy treatment.
Time Frame: 3 Months
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab + GM-CSF
Number analyzed (Participants) | 52
percentage of participants | 69

ADVERSE EVENTS:
Time Frame: Adverse events collected through 8 week treatment period.
Arm/Group | Rituximab + GM-CSF
Serious Adverse Events (participants affected / at risk) | 10/52
Other Adverse Events (participants affected / at risk) | 52/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab + GM-CSF (N=52)
Neutropenia (Blood and lymphatic system disorders) | 8
Pain (General disorders) | 3
Fatigue/weakness (General disorders) | 2
Blurred vision (Eye disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Infusion reaction (Injury, poisoning and procedural complications) | 1
Central Nervous System (CNS) ischemia (Nervous system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab + GM-CSF (N=52)
Allergic Reaction (Immune system disorders) | 1 (1)
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Allergy/Immunology, Other: Mild allergy symptoms (Immune system disorders) | 2 (2)
Blurred Vision (Eye disorders) | 5 (5)
Cardiac General (Cardiac disorders) | 1 (1)
Chest Tightness (Cardiac disorders) | 2 (2)
Confusion (Psychiatric disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 10 (10)
Constitutional Symptoms (General disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dermatology/Skin (Skin and subcutaneous tissue disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 8 (8)
Dizziness (Nervous system disorders) | 9 (9)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9 (9)
Edema, Facial (Skin and subcutaneous tissue disorders) | 4 (4)
Edema: Head And Neck (Skin and subcutaneous tissue disorders) | 2 (2)
Edema: Limb (Skin and subcutaneous tissue disorders) | 5 (5)
Fatigue (General disorders) | 17 (17)
Fever Without Neutropenia (General disorders) | 6 (6)
Flushing (Vascular disorders) | 1 (1)
Gastrointestinal, Other: Gastritis or related symptoms (Gastrointestinal disorders) | 4 (4)
Hemoglobin increased (Investigations) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2)
Hypotension (Metabolism and nutrition disorders) | 1 (1)
Infection (Other) (Infections and infestations) | 1 (1)
Injection Site Reaction (Injury, poisoning and procedural complications) | 7 (7)
Insomnia (Psychiatric disorders) | 1 (1)
Leukocytes Change/Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Memory Impairment (Psychiatric disorders) | 6 (6)
Mental Status (Psychiatric disorders) | 1 (1)
Metabolic/Laboratory, Other: change in blood levels (Metabolism and nutrition disorders) | 1 (1)
Mood Alteration, not interfering with function (Nervous system disorders) | 2 (2)
Mood Alteration (Nervous system disorders) | 1 (1)
Mucositis (Gastrointestinal disorders) | 6 (6)
Musculoskeletal, Other: pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 12 (12)
Neurology (Other) (Nervous system disorders) | 2 (2)
Neuropathy: Motor (Nervous system disorders) | 2 (2)
Neuropathy: Sensory (Nervous system disorders) | 5 (5)
Ocular Surface Discomfort (Eye disorders) | 1 (1)
Ocular/Visual (Eye disorders) | 3 (3)
Pain (Abdomen Nos) (Gastrointestinal disorders) | 2 (2)
Pain (Back) (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain (Bone) (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain (Chest Wall) (General disorders) | 2 (2)
Pain (Chest/Thorax) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pain (Extremity-Limb) (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain (Head/Headache) (General disorders) | 7 (7)
Pain (Muscle) (Musculoskeletal and connective tissue disorders) | 13 (13)
Pain (Neck) (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain (Nos) (General disorders) | 2 (2)
Pain (Other) (General disorders) | 3 (3)
Pain (Scrotum) (Reproductive system and breast disorders) | 1 (1)
Pain (Throat/Pharynx) (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Pulmonary (Other) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash/Desquamation (Skin and subcutaneous tissue disorders) | 2 (2)
Redness Of Eyes (Eye disorders) | 6 (6)
Rigors/Chills (General disorders) | 12 (12)
Sinus Bradycardia (Cardiac disorders) | 1 (1)
Skin Lesion (Skin and subcutaneous tissue disorders) | 1 (1)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Sweating (Skin and subcutaneous tissue disorders) | 3 (3)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Voice Changes (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 6 (6)
Watery Eye (Eye disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes